CLINICAL TRIAL: NCT04963088
Title: Tislelizumab Combined With Anlotinib and Chemotherapy (XELOX) in the Treatment of Advanced Gastric or Gastroesophageal Junction Adenocarcinoma (TALENT): a Single-arm, Open-label Phase I/IIa Trial.
Brief Title: Tislelizumab Combined With Anlotinib and Chemotherapy (XELOX) in the Treatment of Advanced Gastric or Gastroesophageal Junction Adenocarcinoma (TALENT)
Acronym: TALENT
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BGB-A317-ANLO-XELOX GC
Record Dates: First submitted 2021-06-21; First posted 2021-07-15 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2024-04

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — tislelizumab; anlotinib; Oxaliplatin; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TISLELIZUMAB、Anlotinib plus XELOX (Experimental)
  Interventions: Drug: BGB-A317; Drug: Anlotinib; Drug: Oxaliplatin; Drug: Capecitabine

INTERVENTIONS:
Drug: BGB-A317 — Subjects will be treated with BGB A317 200 mg IV on Day 1 during each 21-day cycle. BGB A317 will be administered until disease progression, intolerable toxicity, or treatment discontinuation for any other reason
Drug: Anlotinib — oral administration daily d1-d14, q3w;
Drug: Oxaliplatin — 30 mg/m² IV on Day 1 during each 21-day cycle. during each 21-day cycle
Drug: Capecitabine — 1000 mg/m² orally twice daily (bid) Days 1 through 14 (14 days total) during each 21-day cycle. Capecitabine will be administered until disease progression, intolerable toxicity, or treatment discontinuation for any other reason.

SUMMARY:
This is a Phase 2, multi-cohort study to investigate safety, anti-tumor activity of the monoclonal antibody BGB A317 in combination with Anlotinib and standard chemotherapy as first-line treatment in Gastric, or Gastroesophageal Junction Carcinoma. The study includes a screening (up to 28 days), treatment (until disease progression, intolerable toxicity, or treatment withdrawal for another reason), safety follow-up (up to 30 days following last study drug treatment), and survival follow-up phase.

ELIGIBILITY:
Inclusion Criteria:

1. Able to provide written informed consent and can understand and comply with the requirements of the study
2. Adult patients (≥ 18 years of age or acceptable age according to local regulations, whichever is older) at the time of voluntarily signing informed consent
3. Locally advanced unresectable or metastatic GC or GEJ carcinoma and have histologically confirmed adenocarcinoma
4. At least 1 measurable or non-measurable lesion per RECIST v1.1 as determined by investigator assessment.
5. No previous systemic therapy for locally advanced unresectable or metastatic gastric/GEJ cancer. NOTE: Patients may have received prior neoadjuvant or adjuvant therapy as long as it was completed and have no recurrence or disease progression for at least 6 months.
6. ECOG PS ≤ 1 within 7 days prior to randomization
7. Estimated lifetime is greater than 3 months
8. Adequate organ function as indicated by the following laboratory values ≤ 7 days prior to randomization:

   1. Absolute neutrophil count (ANC) ≥ 1.5 x 109/L, platelets ≥ 100 x 109/L, hemoglobin

      ≥ 90 g/L. NOTE: Patients must not have required a blood transfusion or growth factor support ≤ 14 days before sample collection
   2. Serum creatinine ≤ 1.5 x upper limit of normal (ULN) or estimated Glomerular Filtration Rate ≥ 60 mL/min/1.73 m2. (Appendix 8)
   3. Aspartate transaminase (AST) and alanine aminotransferase (ALT) ≤ 2.5 x ULN
   4. Serum total bilirubin ≤ 1.5 x ULN (total bilirubin must be < 3 x ULN for patients with Gilberts syndrome)
   5. International normalized ratio (INR) or prothrombin time (PT) (or prothrombin time ratio) ≤ 1.5 x ULN unless patient is receiving anticoagulant therapy and PT values are within the intended therapeutic range of the anticoagulant
   6. Activated partial thromboplastin time (aPTT) ≤ 1.5 x ULN
   7. Albumin ≥ 3.0 g/dL or 30 g/liter
9. Weighs more than 40 kg (including 40 kg) or BMI 18.5
10. Females of childbearing potential must have a negative urine or serum pregnancy test within 7 days of randomization and must be willing to use a highly effective method of birth control (Appendix 9) for the duration of the study, and ≥ 120 days after the last dose of tislelizumab or placebo and 180 days after the last dose of chemotherapy.
11. Non-sterile males must be willing to use a highly effective method of birth control (Appendix 9) for the duration of the study and for ≥ 120 days after the last dose of tislelizumab or placebo and 180 days after the last dose of chemotherapy.

Exclusion Criteria:

1. Previous or concurrent other malignant tumors, but cured early tumors, including skin basal cell carcinoma and cervical carcinoma in situ, stage I lung cancer, stage I colorectal cancer.
2. Tumors that do not affect the patient's life in a short period of time as judged by the investigator can be excluded
3. Participation in other drug clinical trials within four weeks;
4. Multiple factors affecting oral medication (such as inability to swallow, chronic diarrhea and intestinal obstruction.
5. History of bleeding, any bleeding event with a severity grade of 3 or higher per CTCAE 5.0 within 4 weeks before screening;
6. Patients with known central nervous system metastasis or history of central nervous system metastasis prior to screening. For patients with clinically suspected central nervous system metastases, CT or MRI must be performed within 28 days before enrollment to rule out central nervous system metastases.
7. Patients with hypertension and uncontrolled by antihypertensive drugs alone (systolic blood pressure > 140 mmHg, diastolic blood pressure > 90 mmHg); Patients with a history of unstable angina pectoris; Patients newly diagnosed as angina pectoris within 3 months before screening or myocardial infarction events within 6 months before screening; Arrhythmias (including QTcF ≥ 450 ms in men, ≥ 470 ms in women requiring long-term use of antiarrhythmic drugs and New York Heart Association Class ≥ II cardiac insufficiency;There are many factors that affect oral drug absorption (such as inability to swallow, nausea and vomiting, upper gastrointestinal obstruction, abnormal physiological function, malabsorption syndrome, etc.), which may affect anlotinib hydrochloride absorbers.
8. Long-term unhealed wound or unhealed fracture;
9. Imaging findings show that the tumor has invaded around important blood vessels or the patient's tumor has a very high possibility of invading important blood vessels during treatment and causing fatal massive hemorrhage as judged by the investigator
10. Patients with abnormal coagulation function and bleeding tendency (the following criteria must be met within 14 days before randomization: INR is within normal range without anticoagulants or has no clinically significant abnormality); patients treated with anticoagulants or vitamin K antagonists such as warfarin, heparin or their analogues; patients with prothrombin time international normalized ratio (INR) ≤ 1.5 are allowed to take low-dose warfarin (1 mg orally, once daily) or low-dose aspirin (the daily dose does not exceed 100 mg) for preventive purposes
11. Arteriovenous thrombotic events occurred within 6 months before screening, such as cerebrovascular accident (including temporary ischemic attack), deep venous thrombosis (except venous thrombosis caused by previous chemotherapy that has been judged by the investigator to have recovered) and pulmonary embolism
12. Urine routine showed urine protein and 24 h urine protein was confirmed to be > 1.0g
13. Previous use of immune targeted therapy drugs;
14. History of immunodeficiency, or other acquired or congenital immunodeficiency diseases, or history of organ transplantation;
15. Patients with infectious pneumonia, pneumonitis, interstitial pneumonia and other conditions requiring corticosteroids;
16. History of severe chronic autoimmune diseases, such as systemic lupus erythematosus; history of inflammatory bowel disease such as ulcerative enteritis, Crohn's disease, irritable bowel syndrome and other chronic diarrheal diseases; history of sarcoidosis or tuberculosis; history of active hepatitis B, C and HIV infection; well-controlled non-serious immune diseases, such as dermatitis, arthritis, psoriasis, etc. Hepatitis B virus < 1000 copies/ml can be detected.
17. Patients with hypersensitivity to human or murine monoclonal antibodies
18. Patients with a history of psychotropic substance abuse and unable to quit or with mental disorders;
19. Pleural or peritoneal effusion with clinical symptoms requiring clinical intervention;
20. Patients who do not follow the doctor's advice, do not take medicine as required, or have insufficient data that can affect the efficacy judgment or safety judgment;
21. Patients with concomitant diseases that, in the judgment of the investigator, seriously jeopardize the patient's safety or affect the patient's completion of the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2021-03-06 (Actual); Primary Completion 2024-03-15 (Actual); Study Completion 2024-03-20 (Actual)

PRIMARY OUTCOMES:
MTD | 6 months
  Maximum tolerated dose
ORR | through study completion, an average of 18 month
  Proportion of patients with reduction in tumor burden of a predefined amount, including complete remission and partial remission

SECONDARY OUTCOMES:
Overall Survival | up to 2 years
  Overall survival was measured from the initiation of chemotherapy to the date of the last follow-up or death.
Progression-free survival | up to 2 years
  he PFS was calculated from the initiation of chemotherapy to the date of disease progression or death.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital with Nanjing Medical University, Nanjing, China

IPD SHARING:
Plan to Share IPD: Undecided